CLINICAL TRIAL: NCT04668105
Title: Effects of Dose Response of Nordic Hamstring Exercise on Muscle Strength, Agility and Speed in Athletes
Brief Title: Dose Response of Nordic Hamstring Exercise on Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00789 SaeedUllah
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Hamstring Injury
Keywords: Agility t test; Eccentric strength; Hamstring injuries; Nordic Hamstring exercises; Single leg Hamstring bridges

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High volume nordic hamstring exercise (Experimental): High volume Nordic hamstring exercise
  Interventions: Other: High volume nordic hamstring exercise
- Low volume Nordic Hamstring exercise (Experimental): Low volume Nordic Hamstring exercise
  Interventions: Other: Low volume nordic hamstring exercise

INTERVENTIONS:
Other: High volume nordic hamstring exercise — To perform Nordic Hamstring Curls, the person will kneel on a pad (for knee comfort) and lower under control, his ankles must be stabilized and kept in a place with the help of a partner, but can also use a moveable object or a loaded barbell can also be used to achieve the stability. The person must then extend his hamstrings in order to lean forward, he should lean forward from the knee and not from the hip. The movement must be kept controlled and slow. The person should go as forward/low as possible but without the help of hands or arms. The only time one can put his hands in front of him is when he can't rely on his legs and then push himself back to starting position and then repeat the procedure again.Group 1 will do the Nordic hamstring exercise with protocol 3 repetitions × 3sets× 3 times for 4 weeks.
  Arms: High volume nordic hamstring exercise
Other: Low volume nordic hamstring exercise — To perform Nordic Hamstring Curls, the person will kneel on a pad (for knee comfort) and lower under control, his ankles must be stabilized and kept in a place with the help of a partner, but can also use a moveable object or a loaded barbell can also be used to achieve the stability. The person must then extend his hamstrings in order to lean forward, he should lean forward from the knee and not from the hip. The movement must be kept controlled and slow. The person should go as forward/low as possible but without the help of hands or arms. The only time one can put his hands in front of him is when he can't rely on his legs and then push himself back to starting position and then repeat the procedure again. Group 2 will do the Nordic hamstring exercise with protocol 3 repetitions × 3 sets × 1 times for 4 weeks.
  Arms: Low volume Nordic Hamstring exercise

SUMMARY:
The aim of this research is to compare the effects of dose response of Nordic hamstring exercise on muscle strength, agility and speed in athletes a randomized controlled trial done at JKD cricket academy and sports centre, Peshawar. The sample size was 34. The subjects were divided in two groups, 17 subjects in Group 1 which will do high volume Nordic hamstring exercise and 17 in Group 2 which will do low volume Nordic hamstring exercise. Study duration was of 6 months. Sampling technique applied was non probability purposive sampling technique. Only 18-30 years athletes with BMI between 18.5-24.5 kg/m2 were included. Tools used in the study are Single leg hamstring bridge (SLHB), Agility t-test, 30-m speed test and muscles size .Data will be analyzed through SPSS 21.

DETAILED DESCRIPTION:
One of the most common injury in sports is the Hamstring injury, as hamstring is very susceptible to tears and strains. Hamstring muscle strain-type injuries are common in sports that involve high degree of speed, power and agility such as sprinters, soccer, basketball, tennis and football. Occurring in both recreational and professional sports, these injuries can result in substantial time lost from sport and commonly recur.

When sprinting, the hamstring muscles of the swing leg function concentrically as hip extensors to quickly swing the thigh back, whereas the same muscle group acts eccentrically as knee flexors to decelerate the forward swing leg. This last action is a probable contributing injury mechanism because of the increased peak hamstring musculotendinous stretch, activation, and active lengthening contraction of the hamstring muscles. The Nordic Hamstring Exercise (NHE) was previously termed the 'Russian hamstring exercise'. This is a partner exercise which can be performed easily on the pitch without special equipment. The NHE involves the player attempting to resist a forward-falling motion from a kneeling position, eccentrically contracting hamstring muscles and thought to replicate hamstring function during terminal swing phase. NHE is a preventive strategy which may reduce the incidence of hamstring injury, medical costs, and personal suffering of the injured player keeping in view the training exposure, training intensity, and compliance to preventive measures. Programs that include the NHE reduce hamstring injuries by up to 51%. The NHE essentially halves the rate of hamstring injuries across multiple sports in different athletes. Even in the face of promising NHE preventive effect shown by previous studies,adoption and implementation of the NHE programs is still low. Evidence show improvement in performance, agility and speed in athletes by NHE training but lowest dose of NHE required to enhance athletes' performance , agility and speed is yet to be found. This study attempts to investigate the lowest dose response of NHE by comparing the effects of high volumes of NHE with low volumes of NHE.

Literature review: Mjølsnes et al first demonstrated that a NHE program performed on the training environment of professional soccer players is more effective in developing maximal eccentric hamstring strength than a comparable program based on hamstring curl machine at the fitness center.

Three large prospective trials (two randomized and one non-randomized) reduced injuries by approximately 70% by implementing the NHE in a team's training regime. The results from the meta-analysis suggested that teams using the NHE (in isolation or as part of a larger injury prevention program) reduced hamstring injury rates up to 51%.

Brooks et al studied the effects of the NHE on the incidence and severity of hamstring strains among 546 professional rugby union players. The NH exercise group had a significantly lower hamstring injury rate and severity than the strengthening and the stretching/ strengthening group.

In a 2020, meta-analyses, positive outcomes were reported on jump performance, repeated sprint ability and agility of athletes after NHE protocol.

A study conducted for 6 weeks concluded that NHE resulted in significant improvements in eccentric strength of hamstrings and performance in 10 m sprinters and also in change of direction speed immediately after the training protocol. These improvements remained even after 3 weeks of detraining.

In a study NHE has shown improvements in strength and dynamic control after 10 weeks of training, a reduction in the maximum peak torque (when approaching full knee extension), and a lower incidence rate of hamstring injuries in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Athletes participating in games for at least 06 months
* BMI 18.5-24.5

Exclusion Criteria:

* Have injuries (prior 6 months) or instability in knee
* Have recently had knee or hip surgery
* Are recovering from injury or surgery involving spine, or neck
* Have ruptured or torn ligaments in knee or ankle, such as Achilles tendon.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Single leg hamstring bridge test | 4th week
  Single leg hamstring bridge (SLHB) is a clinical test for hamstring function used at elite level for the screening programs. To perform this test, person lies on his back with bent knees, hip distance apart, and feet flat on mat stacked under the knees. Extend one leg long towards the ceiling. Squeeze glutes and lift hips off the mat into a bridge. Lower and lift the hips for desired number of repetitions and repeat on other side

SECONDARY OUTCOMES:
Agility t- test | 4th week
  Agility T test is a running test of agility; it involves forward, lateral, and backward movements suitable for a wide range of sports. The subject starts at Cone A. On the command of the timer, the subject sprints to Cone B, and touches the base of the cone with their right hand. They then turn left and shuffle sideways to Cone C, and also touch its base, this time with their left hand. Then shuffling sideways to the right to Cone D and touching the base with their right hand. They then shuffle back to Cone B touching with the left hand, and run backwards to Cone A. The stop watch is stopped as they reach Cone A. We will perform this test for 3 times and will take the best time of the 3 trials.
30-m speed test | 4th week
  30-m Speed test or Sprint test is performed. The time is recorded while the person performs one 30 meters maximum sprint. This test is used to measure the speed and acceleration.
Muscle size | 4th week
  Thigh circumference through anthropometric measuring tape to measure the size of hamstring. The tape will be placed at 5, 10 and 15 cm proximal to superior pole of patella.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- JKD cricket academy and sports Centre,, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Dyk N, Behan FP, Whiteley R. Including the Nordic hamstring exercise in injury prevention programmes halves the rate of hamstring injuries: a systematic review and meta-analysis of 8459 athletes. Br J Sports Med. 2019 Nov;53(21):1362-1370. doi: 10.1136/bjsports-2018-100045. Epub 2019 Feb 26. PMID 30808663
- [Background] Goode AP, Reiman MP, Harris L, DeLisa L, Kauffman A, Beltramo D, Poole C, Ledbetter L, Taylor AB. Eccentric training for prevention of hamstring injuries may depend on intervention compliance: a systematic review and meta-analysis. Br J Sports Med. 2015 Mar;49(6):349-56. doi: 10.1136/bjsports-2014-093466. Epub 2014 Sep 16. PMID 25227125
- [Background] Al Attar WSA, Soomro N, Sinclair PJ, Pappas E, Sanders RH. Effect of Injury Prevention Programs that Include the Nordic Hamstring Exercise on Hamstring Injury Rates in Soccer Players: A Systematic Review and Meta-Analysis. Sports Med. 2017 May;47(5):907-916. doi: 10.1007/s40279-016-0638-2. PMID 27752982
- [Background] Jonhagen S, Nemeth G, Eriksson E. Hamstring injuries in sprinters. The role of concentric and eccentric hamstring muscle strength and flexibility. Am J Sports Med. 1994 Mar-Apr;22(2):262-6. doi: 10.1177/036354659402200218. PMID 8198197
- [Background] Mendiguchia J, Arcos AL, Garrues MA, Myer GD, Yanci J, Idoate F. The use of MRI to evaluate posterior thigh muscle activity and damage during nordic hamstring exercise. J Strength Cond Res. 2013 Dec;27(12):3426-35. doi: 10.1519/JSC.0b013e31828fd3e7. PMID 23524362
- [Background] van der Horst N, Smits DW, Petersen J, Goedhart EA, Backx FJ. The preventive effect of the nordic hamstring exercise on hamstring injuries in amateur soccer players: a randomized controlled trial. Am J Sports Med. 2015 Jun;43(6):1316-23. doi: 10.1177/0363546515574057. Epub 2015 Mar 20. PMID 25794868
- [Background] Krist MR, van Beijsterveldt AM, Backx FJ, de Wit GA. Preventive exercises reduced injury-related costs among adult male amateur soccer players: a cluster-randomised trial. J Physiother. 2013 Mar;59(1):15-23. doi: 10.1016/S1836-9553(13)70142-5. PMID 23419911
- [Background] Junge A, Lamprecht M, Stamm H, Hasler H, Bizzini M, Tschopp M, Reuter H, Wyss H, Chilvers C, Dvorak J. Countrywide campaign to prevent soccer injuries in Swiss amateur players. Am J Sports Med. 2011 Jan;39(1):57-63. doi: 10.1177/0363546510377424. Epub 2010 Oct 17. PMID 20956263
- [Background] Petersen J, Thorborg K, Nielsen MB, Budtz-Jorgensen E, Holmich P. Preventive effect of eccentric training on acute hamstring injuries in men's soccer: a cluster-randomized controlled trial. Am J Sports Med. 2011 Nov;39(11):2296-303. doi: 10.1177/0363546511419277. Epub 2011 Aug 8. PMID 21825112
- [Background] Ribeiro-Alvares JB, Marques VB, Vaz MA, Baroni BM. Four Weeks of Nordic Hamstring Exercise Reduce Muscle Injury Risk Factors in Young Adults. J Strength Cond Res. 2018 May;32(5):1254-1262. doi: 10.1519/JSC.0000000000001975. PMID 28459795